CLINICAL TRIAL: NCT01375179
Title: A Multi-centre, Double-blind, Placebo Controlled, Parallel Group, Proof of Concept Study to Evaluate the Efficacy, Safety and Tolerability of KRP203 in Subjects With Moderately Active Refractory Ulcerative Colitis
Brief Title: Efficacy & Safety in Moderately Active Refractory Ulcerative Colitis Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CKRP203A2201; 2010-019970-33 (EudraCT Number)
Record Dates: First submitted 2011-05-12; First posted 2011-06-17 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2015-05

CONDITIONS: Ulcerative Colitis
Keywords: Inflammatory Bowel disease; Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — KRP-203

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- KRP203 (Experimental): Experimental
  Edit
  Experimental
  Interventions: Drug: KRP203
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo matching KRP203

INTERVENTIONS:
Drug: KRP203
  Arms: KRP203
Drug: Placebo matching KRP203
  Arms: Placebo

SUMMARY:
This study is designed as a proof of concept of KRP203 for induction of remission in ulcerative colitis (UC). The purpose of this study is to evaluate clinical benefit of KRP203 in subjects with moderately active refractory ulcerative colitis.

The study will provide safety and tolerability data in this subject population up to eight weeks of treatment with KRP203. Additionally, this study will evaluate the duration of a clinical response to KRP203 by following up responding subjects for an additional 12 weeks.

DETAILED DESCRIPTION:
This is a multi-centre, double-blind, placebo controlled, parallel group, proof of concept study to evaluate the efficacy, safety and tolerability of KRP203 in subjects with moderately active refractory ulcerative colitis subjects. In total, approximately 72 subjects will be randomized into the study.

After 30 patients have completed the 8 week treatment period with KRP203 or placebo, there will be an interim analysis to determine preliminary efficacy. The study will consist of up to 28 day screening period (day -35 to -8), baseline period (day -7 to day -1), treatment period (day 1 to day 56), follow-up period and study completion.

ELIGIBILITY:
Inclusion Criteria:

* Active disease defined by partial Mayo score and modified Baron score with disease extending at least 25 cm from the anal verge
* Subjects must have inadequately responded or intolerance to 5-ASA therapy

Exclusion Criteria:

* Subjects receiving treatment for UC (other than 5-ASAs and steroids) within the time frame mentioned in protocol
* Past or recent history of significant medical illness and/or clinically significant lab abnormalities including but not limited to hematology, clinical chemistry, urine analysis, ECG abnormalities, HIV, Hepatitis B/C
* Presence or history of underlying metabolic, endocrine, hematologic, pulmonary, ophthalmic, cardiac, blood, renal, hepatic, infectious, psychiatric or any medically unstable condition, as assessed by the primary treating physician which, in the opinion of the investigator, would immunocompromise the subject and/or place the subject at unacceptable risk for participation in a study of an immunomodulatory therapy Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in clinical remission rate | 8 weeks
  Difference between clinical remission rate of subjects on KRP203 versus placebo

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 8 weeks
  Safety and tolerability of KRP203 assessed by the number of subjects with adverse events where KRP203 is given as an oral drug for 8 weeks once a day in ulcerative colitis subjects
Pharmacokinetic properties of KRP203 at steady-state using whole blood samples in patients with ulcerative colitis subjects | 8 weeks
Difference in pharmacokinetic levels | 12 weeks
  To explore the relationship between KRP203 and KRP203-P pharmacokinetic levels and clinical efficacy outcomes such as the partial Mayo score and endoscopic modified Baron Score
Assessment of the pharmacodynamic effect of KRP203 on absolute lymphocyte count and leukocyte subsets in ulcerative colitis subjects | 12 weeks
Change in markers of inflammation | 12 weeks
  Measure of the effect of KRP203 on markers of inflammation, including but not limited to ESR, CRP and fecal calprotectin/ lactoferrin as well as histopathological markers of gut mucosa using biopsy samples in ulcerative colitis subjects

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Belgium (2):
  - Novartis Investigative Site, Ghent
  - Novartis Investigative Site, Leuven
- Germany (3):
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Hamburg
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Sweden (2):
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Switzerland (2):
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Zurich
- United Kingdom (2):
  - Novartis Investigative Site, Oxford, Oxfordshire
  - Novartis Investigative Site, Nottingham